CLINICAL TRIAL: NCT00932581
Title: Investigation of the Psychometric Properties of the Bradykinesia Subscale When Administered Alone Versus as a Component of the Entire Motor Examination Section of the Unified Parkinson's Disease Rating Scale
Brief Title: Bradykinesia Subscale Administered Alone Versus Regular Administration: Psychometric Properties
Acronym: Bravura
Status: Completed | Type: Observational
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Linda Lintz, Clinical Trial Manager, Teva Neuroscience, Inc.
Other Study IDs: PM105
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Movement Disorders; Unified Parkinson's Disease Rating Scale; Short Parkinson's Evaluation Scale; Scales for Outcomes in Parkinson's Disease; Motor Evaluation; Schwab and England activities of daily living; Bradykinesia; psychometrics; order effects; hoehn yahr aging; assessments
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Hypokinesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Full Exam: The first group will receive the full motor examination section in its original order.
  Interventions: Other: Bradykinesia UPDRS Motor Full Examination
- Subscale: The second group will receive the bradykinesia subscale first followed by the remainder of the motor examination section.
  Interventions: Other: Bradykinesia subscale of UPDRS Motor Examination

INTERVENTIONS:
Other: Bradykinesia UPDRS Motor Full Examination — The first group will receive the full motor examination section in its original order.
  Other Names: Experimental group
  Groups: Full Exam
Other: Bradykinesia subscale of UPDRS Motor Examination — The second group will receive the bradykinesia subscale first followed by the remainder of the motor examination section.
  Other Names: Subscale 1, Bradykinesia subscale
  Groups: Subscale

SUMMARY:
The purpose of this study is to examine whether scores on questionnaires that rate how much Parkinson's Disease (PD) has slowed movements of the body differ when the order of the questions are changed. The consistency and accuracy of the questionnaires will also be examined. It is hypothesized that there will not be a difference.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female at least 30 years of age
2. Willing to be assessed using the motor examination section of the UPDRS and the SPES/SCOPA motor evaluation
3. Patients must be willing and able to give written informed consent prior to performing an study procedures
4. Be in the "ON" State (only for patients who fluctuate between "ON" and "OFF" states)

Exclusion Criteria:

1. Absence of bradykinesia at the time of assessment
2. Hoehn and Yahr stage not available from patient's chart or not assessed between 3 and 180 days prior to clinic visit
3. Has received and experimental drug within the last thirty (30) days

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of idiopathic Parkinsons disease (PD) who also presented with bradykinesia and one other cardinal sign at the time of assessment.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Scores on the UPDRS motor evaluation subscale are equivalent. | 4 months

SECONDARY OUTCOMES:
Correlations between the UPDRS motor examination bradykinesis subscale and the remaining UPDRS motor examination items, Hoeh and Yahr stage, Schwab and England scale, and SPES/SCOPA motor evaluation. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Philip Buck, PhD, MPH, Study Director — Teva Neuroscience, Inc.